CLINICAL TRIAL: NCT04444167
Title: An Open-Label Multi-Center Phase Ib/II Study of Anti-PD-1/CTLA-4 Bispecific Antibody AK104 in Combination With Lenvatinib As the First-Line Therapy for Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Anti-PD-1/CTLA-4 Bispecific AK104 Plus Lenvatinib in First-line Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-206
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: VEGF; Anti-PD-1; Tyrosine Kinase Inhibitor (TKI); Anti-CTLA-4
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 and Lenvatinib (Experimental): AK104 6 mg/kg IV every 2 weeks (Q2W) Lenvatinib 12mg weight≥60kg or 8mg weight<60kg,PO QD
  Interventions: Biological: AK104; Drug: Lenvatinib

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 and lenvatinib until disease progression or for a maximum of 24 months
Drug: Lenvatinib — Subjects will receive AK104 and lenvatinib until disease progression for a maximum of 24 months

SUMMARY:
An open-label multi-center phase Ib/II study to evaluate the efficacy and safety of anti-PD-1/CTLA-4 bispecific antibody AK104 plus lenvatinib as the first-line therapy for patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a multi-center, multi-cohort, open-label phase 1b/2 clinical study to evaluate the anti-tumor activity, safety, PK profile, immunogenicity and potential biomarkers of AK104 plus lenvatinib for the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Histologically or cytologically documented hepatocellular carcinoma.
* BCLC stage C, and non-resectable BCLC stage B .
* At least one measurable lesion according to RECIST criteria.
* ECOG of 0 or 1.
* Adequate organ function.
* Estimated life expectancy of ≥3 months.
* For women of childbearing potential: agreement to remain abstinent; For men: agreement to remain abstinent.

Exclusion Criteria:

* Histologically or cytologically documented fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma, etc.
* History of hepatic encephalopathy or liver transplantation.
* Clinical significance of hydrothorax, ascites or pericardial effusion.
* Central nervous system metastases and/or carcinomatous meningitis.
* Any risk of bleeding; severe bleeding tendency or coagulation dysfunction, or under thrombolytic therapy.
* Occurred arteriovenous thromboembolic events within 6 months before the first administration.
* Tumor volume > 50% liver volume; portal vein tumor thrombus or inferior vena cava tumor thrombus.
* Inadequately controlled arterial hypertension.
* Attack of symptomatic congestive heart failure (LVEF<50%); History of congenital long QT syndrome.
* Known presence or history of interstitial lung disease or required hormone treatment interstitial lung disease.
* Severe infections.
* Receipt of any anti-tumor treatment, chemotherapy, targeted therapy, immunotherapy,
* Enrollment of another clinical study within 4 weeks prior to the first administration of study drugs.
* Unable to receive an enhanced CT or MRI scan of the liver.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Number of participants with adverse events (AEs) | the time of informed consent signed through 90 days after the last dose of AK104 and
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Observed concentrations of AK104 | From first dose of AK104 through 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Li Bai, MD, Principal Investigator — Chinese PLA General Hospital; Shunchang Jiao, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Qiao Q, Han C, Ye S, Li J, Shao G, Bai Y, Xu A, Sun M, Wang W, Wu J, Huang M, Song L, Huang L, Liu T, Liu W, Wang ZM, Li B, Xia M, Bai L. The efficacy and safety of cadonilimab combined with lenvatinib for first-line treatment of advanced hepatocellular carcinoma (COMPASSION-08): a phase Ib/II single-arm clinical trial. Front Immunol. 2023 Oct 24;14:1238667. doi: 10.3389/fimmu.2023.1238667. eCollection 2023. PMID 37942328